CLINICAL TRIAL: NCT06171906
Title: Clinical Study of MSCs for Treatment of Poor Graft Function After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Mesenchymal Stem Cells for Treatment of Poor Graft Function After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ShiCang Yu (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Sponsor-Investigator, ShiCang Yu, director of Stem cell and regenerative medicine, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC4PGF
Record Dates: First submitted 2023-11-06; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: MSC
Keywords: allo-HSCT; PGF

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs treatment group (Experimental)
  Interventions: Biological: mesenchymal stromal cells

INTERVENTIONS:
Biological: mesenchymal stromal cells — On the basis of conventional PGF treatment for poor implantation, the enrolled patients were injected with 1×10^6/kg mesenchymal stem cells of cord blood weekly for 4 consecutive weeks

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective approach for treating both benign and malignant blood disorders. It primarily involves high-dose chemotherapy to eliminate tumor cells within the patient's body, as well as to suppress the recipient's hematopoiesis and immune function. The transplantation replaces the recipient's original hematopoietic stem cells (HSCs) with donor-derived HSCs, thereby reconstructing the donor's hematopoietic and immune functions to achieve disease cure.

Poor graft function (PGF) following transplantation, which refers to inadequate engraftment of the transplanted hematopoietic stem cells, is one of the major factors limiting the effectiveness of allo-HSCT. Mesenchymal stromal cells (MSCs), identified within the bone marrow stroma, are a type of non-hematopoietic multipotent stem cells. Several studies, including previous research by our research team, suggest that MSCs can improve the bone marrow hematopoietic microenvironment by secreting various cytokines. This leads to the promotion of hematopoietic stem cell proliferation and differentiation, enhancement of hematopoietic function, and support for hematopoiesis as well as direct or indirect promotion of vascular regeneration in damaged tissues and organs.

Therefore, exploring the efficacy of umbilical cord-derived MSCs in treating poor graft function after allo-HSCT, observing the recovery of blood parameters in patients with poor engraftment, monitoring transplantation-related complications and immune reconstitution, and conducting preliminary investigations into the underlying mechanisms can contribute to the exploration of new clinical techniques for the treatment of PGF following allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Screening patients for allogeneic hematopoietic stem cell transplantation;
2. No gender limit, age ≥18 years old and ≤60 years old;
3. KPS score >60 points, expected survival period >3 months;
4. Those without serious functional damage to important organs throughout the body;
5. The patient has no other contraindications to hematopoietic stem cell transplantation
6. Voluntary test and informed consent.

Exclusion Criteria:

1. Have severe heart, kidney or liver dysfunction;
2. Those combined with other malignant tumors need treatment;
3. There are clinical symptoms of brain dysfunction or severe mental illness and the inability to understand or follow the research protocol;
4. Patients who cannot be guaranteed to complete the necessary treatment plan and follow-up observation;
5. Patients with severe acute allergic reactions;
6. Clinically uncontrolled active infection;
7. Patients who are participating in other clinical trials;
8. Researchers believe that the subject is not suitable for clinical trials for other reasons.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
The Hemogram recovery of patients with poor graft function after treatment | 20~40 days after transplantation
  White blood cells: neutrophil engraftment is defined as neutrophils exceeding 0.5×10^9/L for 3 consecutive days; red blood cells: hemoglobin is not less than 70g/L, and is free of blood transfusion; Platelets: Complete response is defined as platelet count ≥50×10^9/L, continuous for 7 days without platelet transfusion; Partial response (PR) is defined as platelet count (20~50)×10^9/L, continuous Weaning from platelet transfusion at 7 days; no response (NR) is defined as 8 weeks of use at the maximum tolerated dose, platelet count <20×10^9/L or not weaning from platelet transfusion

SECONDARY OUTCOMES:
Infection rate | 20~40 days after transplantation
  Unexpected problems that may occur to the patient or others
graft-versus-host disease | within the initial 30 to 60 days or further
  Graft-versus-host disease (GVHD) is a potentially serious complication of allogeneic stem cell transplantation and reduced-intensity allogeneic stem cell transplantation.
survival rate | 1 year after transplantation
  1-year overall survival and disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Lei Gao, Study Chair — Xinqiao Hospital
Locations (2):
- China (2):
  - Xinqiao Hospital, Chongqing, Shapingba District
  - Second Affiliated Hospital, Army Medical University, PLA, Chongqing

IPD SHARING:
Plan to Share IPD: No
Individual participant data often contains sensitive information, such as personal details, medical history, or financial records. Protecting the privacy and confidentiality of participants is of utmost importance. Sharing such data without proper safeguards could violate privacy regulations or ethical considerations.

REFERENCES:
- [Background] Kong Y, Song Y, Tang FF, Zhao HY, Chen YH, Han W, Yan CH, Wang Y, Zhang XH, Xu LP, Huang XJ. N-acetyl-L-cysteine improves mesenchymal stem cell function in prolonged isolated thrombocytopenia post-allotransplant. Br J Haematol. 2018 Mar;180(6):863-878. doi: 10.1111/bjh.15119. Epub 2018 Feb 2. PMID 29392716
- [Background] Michalicka M, Boisjoli G, Jahan S, Hovey O, Doxtator E, Abu-Khader A, Pasha R, Pineault N. Human Bone Marrow Mesenchymal Stromal Cell-Derived Osteoblasts Promote the Expansion of Hematopoietic Progenitors Through Beta-Catenin and Notch Signaling Pathways. Stem Cells Dev. 2017 Dec 15;26(24):1735-1748. doi: 10.1089/scd.2017.0133. Epub 2017 Nov 27. PMID 29050516

DOCUMENTS (1):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT06171906/Prot_000.pdf